CLINICAL TRIAL: NCT04953572
Title: Autologous Peripheral Blood Mesenchymal Stem Cell Transplantation for Repair of Degree IV Local Cartilage Injury of Knee Joint
Brief Title: Treatment of Cartilage Defects With Peripheral Blood Stem Cells
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Inner Mongolia People's Hospital (Other); Hebei Medical University Third Hospital (Other); Tianjin Hospital (Other)
Responsible Party: Principal Investigator, Yu Jiakuo, Chief physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PekingUTH001
Record Dates: First submitted 2021-06-15; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Cartilage Injury
MeSH Terms: interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- test group (Experimental): Patients in the test group received autologous peripheral blood mesenchymal stem cell therapy
  Interventions: Genetic: autologous peripheral blood mesenchymal stem cell
- control group 1 (Active Comparator): Patients in the control group 1 received microfracture surgical treatment
  Interventions: Procedure: Microfracture
- control group 2 (Active Comparator): Patients in the control group 2 received microfracture combined with surgical treatment of collagen membrane
  Interventions: Combination Product: Microfracture + collagen membrane
- control group 3 (Active Comparator): Patients in the control group 3 received autologous osteochondral transplantation
  Interventions: Procedure: Autologous osteochondral transplantation

INTERVENTIONS:
Genetic: autologous peripheral blood mesenchymal stem cell — Transplantation of autologous peripheral blood mesenchymal stem cell
  Arms: test group
Procedure: Microfracture — Microfracture
  Arms: control group 1
Combination Product: Microfracture + collagen membrane — Microfracture plus collagen membrane transplantation
  Arms: control group 2
Procedure: Autologous osteochondral transplantation — Autologous osteochondral transplantation
  Arms: control group 3

SUMMARY:
Knee joint cartilage cells metabolize slowly, and it is difficult to repair themselves after injury. Any knee joint trauma or the progression of osteoarthritis may lead to the progression of cartilage or osteochondral defects. Compared with bone marrow mesenchymal stem cells (MSCs), peripheral blood MSCs have better chondrogenic differentiation ability. At the same time, the mobilization of peripheral blood MSCs and the advancement of extraction technology also make it feasible to treat osteochondral damage by using peripheral blood MSCs. The purpose of this study is to evaluate the therapeutic effect of surgical transplantation of autologous peripheral blood MSCs to repair knee joint Ⅳ-degree localized cartilage injury, and to explore a new treatment for osteochondral defects based on the foundation of the research group's previous research.

DETAILED DESCRIPTION:
1. Explore the clinical efficacy of autologous peripheral blood mesenchymal stem cell transplantation in the treatment of osteochondral defects
2. Exploring the characteristics of cartilage regeneration in autologous peripheral blood mesenchymal stem cell transplantation

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 18 and under 60, regardless of gender.
2. Symptoms, signs and imaging changes are consistent with knee joint limitations IV cartilage defect or patella chondromalacia, patellofemoral joint cartilage injury, mild to moderate knee osteoarthritis.
3. Other treatments are ineffective.
4. No treatment for other knee cartilage defects during the specified period of the test.
5. The subject must be able to communicate well with the researcher and comply with the research requirements, and must give written, signed and dated informed consent before conducting any research-related activities. All relevant legal representatives will also sign a written research agreement in accordance with local laws and regulations.

Exclusion Criteria:

1. The diameter of the cartilage defect in the patient is less than 5mm.
2. Grade Ⅲ and Ⅳ knee joint OA.
3. The patient's symptoms and signs are not closely related to the cartilage defect area.
4. Suffering from concomitant inflammatory diseases (such as rheumatoid arthritis), osteochondrotis dissecans, sepsis, osteonecrosis, and various tumor diseases in the past; in the past three months, there was in the joint cavity of the affected knee History of injection.
5. Suffer from the underlying medical conditions (including but not limited to metabolism, hematology, kidney, liver, lung, nerve , Endocrine, heart, infection, or gastrointestinal tract); currently suffering from a serious progressive or uncontrolled disease that is not suitable for the test or puts it at high risk, including the researchers belief that it will prevent the subject from following the protocol or completing the study according to the protocol Any medical or psychiatric condition of
6. Being infected with human immunodeficiency virus (HIV), infectious hepatitis B or hepatitis C or corresponding medical history.
7. Suffer from a progressive infection or malignant disease, and be able to produce chest X-ray, computed tomography (CT scan) or MRI evidence within 12 weeks before screening, and be evaluated and confirmed by a qualified physician.
8. Active systemic infections (except colds) or any other infections that will recur regularly in the previous two weeks.
9. There is a history of chronic or recurrent infectious diseases, or evidence of tuberculosis infection that was judged to be positive at the time of screening. Subjects who have obtained positive or uncertain results can participate in the study if they undergo a comprehensive tuberculosis examination (according to local practice/guidelines) within 12 weeks before baseline and finally prove that there is no evidence of active tuberculosis. If the presence of latent tuberculosis is confirmed, treatment must be initiated and maintained in accordance with local or national guidelines before the baseline.
10. History of lymphoproliferative disease, or any known malignant tumor, or history of malignant tumor of any organ system in the past 5 years (Bowen's disease, basal cell carcinoma, or actinic keratosis after treatment and no evidence of recurrence in the past 12 weeks Except for diseases; except for excised cervical carcinoma in situ or non-invasive malignant colon polyps).
11. Suffer from medical problems at the same time, including but not limited to the following:
12. Uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥95mmHg), congestive heart failure (New York Heart Association status classification III or IV).
13. Subjects whose serum creatinine level exceeds 2.0 mg/dl (176.8 μmol/L).
14. Total white blood cell (WBC) count at screening <2500/μL, or platelet <100000/μL or neutrophil <1500/μL or hemoglobin <8.5 g/dL.
15. For pregnant or lactating women, pregnancy is defined as the state of a woman after conception until the termination of pregnancy, which is confirmed by the positive result of the hCG laboratory test.
16. Women with childbearing potential are defined as all women who are physiologically able to become pregnant, unless they use effective contraceptive methods during the entire study treatment administration period.
17. In the six months before the baseline, there is a history of alcohol or drug abuse or evidence of ongoing abuse.
18. A history of allergies to the components of the therapeutic drugs used.
19. The returning visitors cannot be tracked in time.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 252 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Magnetic Resonance Imaging in the 6th month after surgery | 6 months after sugery
  Magnetic Resonance Imaging，including T2-mapping sequence, to evaluate the magnetic resonance observation of cartilage repair tissue (MOCART) score of cartilage regeneration in the knee articular cartilage defect area at 6 months after sugery. The MOCART score ranges from 0 to 100 points, the higher the score, the better the repair effect.
Magnetic Resonance Imaging in the 12th month after surgery | 12 months after sugery
  Magnetic Resonance Imaging，including T2-mapping sequence, to evaluate the MOCART score of cartilage regeneration in the knee articular cartilage defect area at 12 months after sugery
Magnetic Resonance Imaging in the 24th month after surgery | 24 months after sugery
  Magnetic Resonance Imaging，including T2-mapping sequence, to evaluate the MOCART score of cartilage regeneration in the knee articular cartilage defect area at 24 months after sugery

SECONDARY OUTCOMES:
The Western Ontario and McMaster Universities (WOMAC) Osteoarthritis Index | 3, 6, 12, 18 and 24 months after sugery
  The higher the WOMAC osteoarthritis index, the more severe the OA. Evaluate the severity of OA according to the following criteria: less than 80 is mild, 80-120 is moderate, and greater than 120 is severe.
International knee documentation committee (IKDC) Knee Joint Score Sheet | 3, 6, 12, 18 and 24 months after sugery
  IKDC is an internationally recognized score sheet for comprehensive evaluation of the subjective symptoms and objective signs of the knee joint system.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-kuo Yu, Prof., Study Chair — Peking University Third Hospital
Locations (1):
- Institute of Sports Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No